CLINICAL TRIAL: NCT00895271
Title: Establishing Fibroblast-derived Cell Lines From Skin/Tissue Biopsies of Patients With Immunodeficiency or Immunodysregulation Disorders
Brief Title: Establishing Fibroblast-Derived Cell Lines From Skin Biopsies of Patients With Immunodeficiency or Immunodysregulation Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090133; 09-I-0133
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Primary Immunodeficiency; DOCK8; Virus Susceptibility
Keywords: FIBROBLAST; Skin Biopsy; Innate Immunity; Induced Pluripotent; Natural History; Primary Immunodeficiency; Immunodysregulation; Common Variable Immunodeficiency; Severe Combined Immunodeficiency; Healthy Volunteer; HV
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; Severe Combined Immunodeficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Up to 50 subjects as healthy controls
- Immunodeficiency: Up to 150 subjects with poorly defined, rare inherited immunodeficiency or immunodysregulation disorders

SUMMARY:
Background:

* National Institutes of Health (NIH) researchers have been studying immune cells (white blood cells) to better understand how the human body s defense system works and adjusts or regulates itself, and how changes in this system can make a person sick.
* To study the cells of patients who have problems with their immune systems, researchers would like to collect samples of skin cells from patients with immune system disorders and compare them with skin cells taken from healthy volunteers. By studying these cells, researchers hope to determine whether these cells can be modified to create a new kind of personalized gene therapy that would attempt to cure immune diseases in the future.

Objectives:

* To obtain skin cells from patients with immune system disorders and from healthy volunteers for research and comparison purposes.

Eligibility:

* Patients between the ages of 2 and 85 who have immune system disorders.
* Healthy volunteers between the ages of 18 and 85.
* Both groups will be selected from the eligible participants of existing NIH studies into immune system disorders.

Design:

* Researchers may take up to two biopsies from participants arms, legs, abdomen, or back.
* The biopsy site will be numbed with local anesthetic and cleaned before the sample is taken.
* The punch skin biopsy needle will be inserted into the skin and rotated to remove a small circle of skin (approximately 1/4 to 3/8 of an inch across). The area will be closed with bandages or stitches, and then covered with a dressing. Any stitches will be removed in 7 to 10 days.
* Tissue samples collected in the study will be stored for future research.

DETAILED DESCRIPTION:
This protocol is designed as an adjunct to other National Institutes of Health (NIH) IRB approved protocols that allow for genetic testing, which may include those that are screening protocols for patients with rare primary immunodeficiency or immunodysregulation disorders. Patients deemed of sufficient research interest after review of outside medical records, clinical evaluation, and testing, may be invited to participate in this study. Healthy volunteers and relatives of patients will also be invited to participate as a source of control samples for research testing. After consent and enrollment into this study, skin punch biopsies will be obtained to establish dermal fibroblast cell lines for research studies directed at understanding the genetic and biochemical bases of these diseases. Cell lines will also be used to investigate the utility of induced pluripotent stem cells (iPS) for lymphocyte derivation and targeted gene correction. The nasal epithelial scrapings will be used for research purposes to grow out primary nasal respiratory epithelial cell lines. These cell lines will be used for functional studies by testing virus replication in them. These functional studies will allow us to identify new primary immunodeficiencies that may present primarily as recurrent or persistent lower respiratory tract virus infections. Results with the potential to impact medical care will be relayed to the referring physicians and where applicable patients will be referred to other appropriate NIH protocols for additional clinical evaluation and treatment.

The study will enroll up to 200 patients and healthy volunteers over the next 27 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients:

1. To be enrolled in this study, a patient must be >=2 years of age but not >85 years of age,
2. have a known diagnosis of primary immunodeficiency or immunodysregulation (or be a blood relative of such as patient),
3. be concurrently enrolled on an NIH IRB approved NIAID protocol that includes genetic testing for disease of the immune system, such as but not limited to 05-I-0213 or 06-I-0015

Patient Relative: To be enrolled in this study, a patient relative must be:

1. A biological relative of a participant being studied under this protocol. Relatives may be biological mother, father, sibling, children, grandparents, aunts, uncles and first cousins.

   a. A minor relative of the proban participant must demonstrate that they are asymptomatic carriers or are at risk for the disease
2. be concurrently enrolled on an NIH IRB approved protocol that includes genetic testing for disease of the immune system, such as but not limited to 05-I-0213 or 06-I-0015.
3. Greater than or equal to 8 years of age but not greater than 85 years of age,

Healthy Volunteers:

To be enrolled in this study, a normal volunteer must fulfill all of the following criteria:

1. Be enrolled on protocol 05-I-0213.
2. Be a healthy adult of either sex and between ages of 18 years and 85 years

EXCLUSION CRITERIA:

Patients or the Patient Relative are not eligible to be in this trial if::

1. Platelet count less than 20,000/microL
2. The individual is hemodynamically unstable because of acute bleeding.
3. Any condition that, in the investigator s opinion, places the patient at undue risk by participating in the study or limits the utility of the specimen to be obtained.
4. For Nasal Scraping: a history of turbinectomy or significant nasal pathology that would preclude obtaining mucosal scrape biopsies.

A Healthy Volunteer is not eligible to be in this trial if they:

1. Areless than 18 years old or older than 85 years
2. Weighs less than 110 pounds
3. Are pregnant or breastfeeding
4. Are receiving a chemotherapeutic agent(s) or has a malignancy
5. Cannot avoid taking aspirin or non-steroidal anti-inflammatory medications during the 7 days preceding skin biopsy
6. Have history of heart, lung, kidney disease, bleeding disorders, diabetes mellitus, chronic peripheral arterial or venous insufficiency, chronic diffuse skin conditions without uninvolved areas suitable for skin biopsy, poor skin healing, or keloid formation.
7. Have been diagnosed as having viral hepatitis (B or C), human immunodeficiency virus (HIV), or a carrier for methicillin-resistant Staphylococcus aureus (MRSA)
8. Hemoglobin measurement is less than 12.0 g/dL
9. Platelet count less than 150,000/(micro)L
10. PT greater than 15.0 seconds or PTT greater than 40 seconds
11. Have a history of intravenous injection drug use or of engaging in high-risk activities for exposure to the acquired immunodeficiency syndrome (AIDS) virus.

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Up to 150 patients with poorly defined, rare inherited immunodeficiency or immunodysregulation disorders, and up to 50 healthy volunteers as controls. Patients and healthy volunteers, who are first evaluated under another NIAID protocol (such as 05-I-0213 or 06-I-0015) and others, may be offered the opportunity to participate in this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-06-10 (Actual)

PRIMARY OUTCOMES:
Generate fibroblast, dermal, or other skin-resident cell lines | Over the lifetime of the study
  Obtain skin punch biopsies to generate fibroblast, dermal, or other skin-resident cell lines in patients who previously underwent HSCT. Cells may also be used for somatic cell hybridization, cell complementation, assessing fibroblast-specific innate immune responses, or other genetic techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Su, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There isn't any data generated on this study that is relevant or shareable to any individual participant. Data obtained from iPS line growth is not medically actionable and therefor will not be reported back or shared with the participant.

REFERENCES:
- [Background] Hernandez N, Melki I, Jing H, Habib T, Huang SSY, Danielson J, Kula T, Drutman S, Belkaya S, Rattina V, Lorenzo-Diaz L, Boulai A, Rose Y, Kitabayashi N, Rodero MP, Dumaine C, Blanche S, Lebras MN, Leung MC, Mathew LS, Boisson B, Zhang SY, Boisson-Dupuis S, Giliani S, Chaussabel D, Notarangelo LD, Elledge SJ, Ciancanelli MJ, Abel L, Zhang Q, Marr N, Crow YJ, Su HC, Casanova JL. Life-threatening influenza pneumonitis in a child with inherited IRF9 deficiency. J Exp Med. 2018 Oct 1;215(10):2567-2585. doi: 10.1084/jem.20180628. Epub 2018 Aug 24. PMID 30143481
- [Background] Lamborn IT, Jing H, Zhang Y, Drutman SB, Abbott JK, Munir S, Bade S, Murdock HM, Santos CP, Brock LG, Masutani E, Fordjour EY, McElwee JJ, Hughes JD, Nichols DP, Belkadi A, Oler AJ, Happel CS, Matthews HF, Abel L, Collins PL, Subbarao K, Gelfand EW, Ciancanelli MJ, Casanova JL, Su HC. Recurrent rhinovirus infections in a child with inherited MDA5 deficiency. J Exp Med. 2017 Jul 3;214(7):1949-1972. doi: 10.1084/jem.20161759. Epub 2017 Jun 12. PMID 28606988
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-I-0133.html